CLINICAL TRIAL: NCT06877273
Title: CIRCuiTS MS: Improving Cognitive Recovery in Multiple Sclerosis
Brief Title: Improving Cognitive Recovery in Multiple Sclerosis
Acronym: CIRCuiTS-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 348879
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive rehabilitation; cognitive training; cognitive remediation; thinking skills; randomised controlled trial; feasibility; acceptability; metacognition; cognitive remediation therapy; cognitive dysfunction; cognitive function
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups:
  1. Immediate Treatment Group: Participants will start the cognitive remediation program immediately.
  2. Delayed Treatment Group: Participants will be placed on a waitlist and receive the program after 14 weeks
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): Participants will start the cognitive remediation program immediately after recruitment. Outcome measures will be taken before treatment (week 1), immediately after treatment (week 14), and at 14 weeks after end of treatment (week 27).
  Interventions: Behavioral: CIRCuiTS-MS
- Delayed Treatment Group (Experimental): Participants will start the cognitive remediation program after being on a waitlist for 13 weeks. Outcome measures will be taken when added to the waitlist (week 1), before treatment (week 14), and immediately after treatment (week 27).
  Interventions: Behavioral: CIRCuiTS-MS

INTERVENTIONS:
Behavioral: CIRCuiTS-MS — The intervention is a blended treatment combining therapist support with carrying out tasks in CIRCuiTS™ digital cognitive remediation software. This software provides opportunities to practice a range of cognitive tasks and adaptively adjusts task difficulty. CIRCuiTS™ is much used in psychosis. Based on collaborative workshops with people with MS, participants for this trial will be asked to attend two 1-hour therapy sessions (in person or on MS Teams) and 1 hour of independent tasks each week for 12 weeks. Participants with reduced ability to operate a mouse quickly or dexterously will be offered a modified programme omitting tasks that require these abilities. The therapist will be an Assistant Psychologist trained in CIRCuiTS™ delivery and in appropriate adjustments to the needs of people with MS. They will follow a manualised template and will receive weekly supervision from an experienced clinical psychologist.

SUMMARY:
This study aims to find out whether an adapted version of an existing cognitive rehabilitation program, CIRCuiTS (https://www.circuitstherapyinfo.com), can be used to improve everyday thinking skills for people with Multiple Sclerosis (MS). People living with MS have worked with the study's researchers to adapt CIRCuiTS to meet their needs. They shared the thinking challenges they experience and suggested changes to the program's content and how it is delivered. This study will test whether this adapted version can be delivered practically to people with MS in a trial setting and explore its potential benefits. The findings will help plan a larger trial testing how effective CIRCuiTS is in helping people with MS.

Twenty-four people with MS will take part in this pilot trial. Each person will be randomly assigned to start the program either right away or after a 13-week wait. The therapy program involves up to 36 hours of therapist-led and independent sessions over 12 weeks in which the participant builds thinking skills through developing personal strategies for carrying out digital versions of tasks they find challenging. The practicality of delivering the program to people with MS will be judged based on whether problems arise in the trial, such as not being able to recruit enough people or participants not liking it. To explore its potential benefits, the study will check for improvements in progress toward personal goals, thinking abilities, emotional well-being, chronic tiredness, and daily living skills after the therapy.

If delivering CIRCuiTS to people with MS is found to be both practical and acceptable to participants, the findings of this trial will be used to design a larger-scale trial of its effectiveness. Ultimately, the goal of this project is to improve the quality of life of people living with cognitive difficulties related to MS.

DETAILED DESCRIPTION:
Objectives

The primary goal of this study is to assess the practical aspects of the research to determine whether a larger, fully-scale trial will be viable and acceptable. A feasibility decision will be reached by judging whether a suite of "Go"/"No-Go" thresholds associated with the primary outcome measures have been passed. Additionally, acceptability will be explored through qualitative analysis of participant exit interviews.

The secondary goal is to explore the potential that a larger trial will show that the program helps people with MS in meaningful ways.

Specifically, the study will examine whether the cognitive remediation program:

1. Helps participants meet their personal goals
2. Improves participants' cognitive function (how they think and think about thinking)
3. Improves participants' mood (specifically feelings of anxiety and depression, which are common in people with MS)
4. Helps reduce the severe fatigue that many people with MS experience
5. Affects participants' ability to carry out everyday activities, such as managing tasks at home, working, and engaging in social and leisure activities.

These factors will be evaluated through assessing change in the secondary outcome measures after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of Multiple Sclerosis (MS), as verified by a healthcare provider.
* Participants should be in a relatively stable phase of their condition, not experiencing a severe relapse or acute health crisis at the time of the study.
* Participants must have sufficient cognitive abilities to engage in therapy sessions, meaning they can follow instructions and perform the cognitive tasks required during the remediation program.
* Participants must be able to effectively communicate in English, both verbally and in writing, to interact with therapists and complete assessments.
* Participants must be adults aged 18 years or older.
* Participants should have personal experience with cognitive challenges related to MS, such as problems with memory, attention, or problem-solving.
* Participants must be willing and able to commit to attending all therapy sessions over the 12-week period, as well as attending assessments and completing any required homework or independent sessions.
* Participants must provide informed consent, demonstrating that they understand the purpose of the therapy trial and are willing to engage in the course of cognitive remediation.
* Participants must have access to a computer (laptop or desktop) for at least one hour per week during the treatment period (12 weeks).

Exclusion Criteria:

* Individuals who are currently receiving cognitive remediation or a similar intervention.
* Individuals with high levels of depression, indicated by a score greater than 9 on the Patient Health Questionnaire-9 (PHQ-9).
* Individuals with active suicidal ideation, indicated by a score greater than 0 on question 9 of the PHQ-9.
* Individuals with a diagnosis of a psychotic disorder or bipolar disorder.
* Physical disabilities that severely limit the individual's ability to attend therapy sessions or engage with the cognitive tasks (whether in-person or online) may lead to exclusion if suitable adaptations cannot be made.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Until the end of the study, estimated 15 months
  Percentage of planned sample size recruited
Ethnic enrolment diversity | Until the end of the study, estimated 15 months
  Percentage of sample belonging to the most common ethnicity
Gender enrolment diversity | Until the end of the study, estimated 15 months
  Difference in the percentages of recruited participants identifying as male and female
Completion rate | Until the end of the study, estimated 15 months
  Percentage of participants completing week 27 measures
Midpoint retention | Until the end of the study, estimated 15 months
  Percentage of participants completing week 14 measures
Dropout | Until the end of the study, estimated 15 months
  Percentage of enrolled participants who drop out
Serious adverse events | Until the end of the study, estimated 15 months
  Number of serious adverse events reported
Manageability of adverse events | Until the end of the study, estimated 15 months
  Number of adverse events that cause the study to be halted
Data completeness | Until the end of the study, estimated 15 months
  Percentage outcome data complete
Specific measure completeness | Until the end of the study, estimated 15 months
  Percentage outcome data complete per measure
Operational feasibility | Until the end of the study, estimated 15 months
  Number of significant operational issues that cannot be resolved
Adherence: Therapy | Until the end of the study, estimated 15 months
  Percentage participants attending ≥ 70% of therapy sessions
Adherence: Independent sessions | Until the end of the study, estimated 15 months
  Percentage participants attending ≥ 40% of therapy sessions
Specific measure acceptability | Until the end of the study, estimated 15 months
  Percentage of participants who provide answers to demographic/medical background questions
Program acceptability | Until the end of the study, estimated 15 months
  Mean score on the general acceptability item of the Theoretical Framework of Acceptability Questionnaire

SECONDARY OUTCOMES:
Goal Attainment Scale | From goal setting in week 1 to week 27
  A personalised measure used to assess the extent to which patient-specific goals are achieved during therapy. Goals are collaboratively set between the therapist and patient, and the level of attainment is rated on a scale typically ranging from -2 (much less than expected outcome) to +2 (much more than expected outcome).
Measure of Insight into Cognition | From baseline assessment at week 1 to week 27
  A self-report questionnaire designed to assess an individual's awareness and understanding of their cognitive abilities and deficits. It is particularly useful in clinical settings where cognitive impairments are common, such as in MS. The MIC consists of a series of statements that participants rate based on their perception of their cognitive functions. Each item is rated on a Likert scale, ranging from 1 to 5, from strongly agree to strongly disagree. The total score is the sum or average of the scores for the items. Higher scores indicate greater insight into one's cognitive abilities and deficits.
Brief International Cognitive Assessment for Multiple Sclerosis | From baseline assessment at week 1 to week 27
  Designed for rapid assessment of neuropsychological abilities commonly affected in MS. Comprises:
  The Symbol Digit Modalities Test, measuring processing speed and attention. The participant is asked to orally identify the digits associated with test symbols within a key. It is scored on the number of digits correctly identified within 90 seconds.
  Tasks 1-3 of the Brief Visuospatial Memory Test, measuring immediate visual recall. The participant inspects an array of 6 abstract geometric figures during three 10-second learning trials and then draws the array from memory. Higher scores are awarded for more accurate figure reproduction and positioning.
  Tasks 1-5 of the California Verbal Learning Test-Second Edition, measuring verbal working memory. The rater reads a 16-item word list aloud five times to the participant, who is then required to recall as many as possible.
Digit Span | From baseline assessment at week 1 to week 27
  This subtest from the Wechsler Adult Intelligence Scale Version 4 will be administered because it is a widely used measure of attention and working memory that does not show strong correlations with the California Verbal Learning Test. The participants is required to repeat sequences of digits, proceeding to longer sequences if correct, then repeat sequences backwards and in numerical order.
Controlled Oral Word Association Test | From baseline assessment at week 1 to week 27
  A widely used neuropsychological assessment tool designed to measure verbal fluency, a component of executive function. It assesses the ability to generate words according to specific phonemic and semantic criteria within a limited time frame. The COWAT is commonly used in the diagnosis and evaluation of various neurological and psychiatric conditions. To measure phonemic fluency, participants are asked to produce as many words as possible that begin with a specific letter (usually F, A, and S) within 60 seconds for each letter. To measure semantic fluency, participants are asked to produce as many words as possible within a category (e.g., animals) within 60 seconds. The number of correct words generated in each category (phonemic and semantic) is counted. Repetitions, proper nouns, and variations of the same word are not included in the score. Errors will also be analysed, such as repetitions or rule violations, providing additional insights into cognitive function.
Patient Health Questionnaire-9 | From baseline assessment at week 1 to week 27
  A widely used self-administered tool for screening, diagnosing, monitoring, and measuring the severity of depression. It is based on the diagnostic criteria for major depressive disorder outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). The PHQ-9 consists of 9 items, each corresponding to one of the DSM-IV criteria for depression. Each item is rated on a 4-point Likert scale based on the frequency of symptoms over the past two weeks. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Generalised Anxiety Disorder Scale | From baseline assessment at week 1 to week 27
  A brief, self-report screening tool commonly used in clinical and research settings to assess the severity of generalised anxiety disorder (GAD) symptoms. The GAD-7 provides an efficient way to identify GAD symptoms and track their severity over time. The GAD-7 contains 7 questions that evaluate the frequency of core anxiety symptoms over the past two weeks. Total scores range from 0 to 21, with higher scores indicating greater anxiety severity.
Fatigue Severity Scale | From baseline assessment at week 1 to week 27
  A self-report questionnaire designed to assess the impact of fatigue on a person's daily life. It is widely used in clinical and research settings to evaluate fatigue in various conditions, including multiple sclerosis (MS). The FSS consists of 9 statements related to the severity and impact of fatigue. Each item is rated on a 7-point Likert scale. The total score is the average of the scores for the 9 items, resulting in a score range from 1 to 7. Higher scores indicate greater fatigue severity and impact.
Work and Social Adjustment Scale | From baseline assessment at week 1 to week 27
  A self-report questionnaire designed to assess the impact of a person's mental health on their daily functioning. It is widely used in both clinical and research settings to gauge the extent to which psychological problems interfere with a person's ability to perform various life roles. The WSAS consists of 5 items, corresponding to five domains of daily functioning: work, home management, social leisure activities, private leisure activities, and family and relationships. Each item is rated on an 8-point Likert scale from 0 (not at all impaired) to 8 (severely impaired). The total score is the sum of the ratings for the five items, resulting in a score range from 0 to 40. Higher scores indicate greater impairment. A total score of 20 or above suggests significant functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Simblett, PhD, Principal Investigator — King's College London; Til Wykes, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, East of England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified text-based participant data and a data dictionary describing the data types collected will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available from the end of analysis (anticipated September 2026).
Access Criteria: Data and supporting information will be shared upon application to the listed study team.

REFERENCES:
- See also: Website introducing the CIRCuiTS intervention — https://www.circuitstherapyinfo.com